CLINICAL TRIAL: NCT00361621
Title: Phase II Study of CHOP/Rituxan Plus VELCADE in Mediastinal Large B-cell Lymphoma
Brief Title: Ph II CHOP+Velcade in Mediastinal LBCL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Closed due to slow accrual
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Ann S. LaCasce, MD, Assistant Professor of Medicine, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-012; X05194
Record Dates: First submitted 2006-08-07; First posted 2006-08-08 (Estimated); Last update posted 2012-12-03 (Estimated); Status verified 2009-10

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: VELCADE
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Bortezomib; Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone; Radiotherapy

INTERVENTIONS:
Drug: bortezomib — Given intravenously on day 1 and day 4 of a 21-day cycle for 6 cycles
  Other Names: Velcade
Drug: Rituximab — Given intravenously on day 1 of a 21-day cycle for 6 cycles
Drug: Cyclophosphamide — Given intravenously on day 1 of a 21-day cycle for 6 cycles
Drug: Doxorubicin — Given intravenously on day 1 of a 21-day cycle for 6 cycles
Drug: Vincristine — Given intravenously on day 1 of a 21-day cycle for 6 cycles
Drug: Prednisone — Taken orally on days 2, 3, 4 and 5 or a 21-day cycle for 6 cycles
Radiation: Radiation therapy — After 6 cycles of chemotherapy there will be 3 weeks of radiation therapy

SUMMARY:
The main purpose of this study is to begin to collect information and try to learn whether or not VELCADE, when added to standard chemotherapy with CHOP/Rituxan, works in treating patients mediastinal large B-cell lymphoma. Recent research has shown that this type of lymphoma shares features with Hodgkin's lymphoma, including the importance of a particular pathway in the tumor cells called the NF-kB pathway. VELCADE works in part by blocking this pathway.

DETAILED DESCRIPTION:
* This is a single arm phase 2 study of CHOP/Rituxan plus VELCADE followed by involved field radiotherapy designed to evaluate the complete response to chemotherapy as determined by PET scan following six cycles of therapy. One cycle equals 21 days.
* For each cycle, on Day 1, the patient will receive VELCADE intravenously, followed by rituxan, and then followed by CHOP chemotherapy. Before receiving these drugs, the patient will be given standard medications (Tylenol, Benadryl) to help minimize side effects. They will also continue to take prednisone by mouth on days 2, 3, 4, and 5. On Day 4, the patient will receive another dose of VELCADE.
* Before the beginning of every cycle of study treatment, the following will be performed: Medical history; physical examination; and routine blood tests. After the 3rd and 6th cycle of study treatment, the patient will have tests to monitor the status of their disease. These include PET scan, CT scans, and standard blood tests.
* After 6 cycles of chemotherapy, approximately 3 weeks of radiation therapy will begin. One month after completing radiation therapy, the patient will return to the clinic for a physical exam and blood tests. One month later, the following evaluations will occur: PET and CT scans; medical history; physical exam; routine blood tests.
* There will be follow-up visits every 3 months for two years after the study treatment is completed.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
* Female subject is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control (ie, a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study.
* Male subject agrees to use an acceptable method for contraception for the duration of the study.
* Histologic Documentation: Histologically confirmed Primary Mediastinal Large B-cell Lymphoma with confirmatory immunoperoxidase stains including TRAF-1, and nuclear c-rel. All cases must be reviewed at Brigham and Women's Hospital.
* Previously untreated patients with the exception of limited radiotherapy or steroids for SVC syndrome
* Age > 18 years of age
* Measurable Disease defined as lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥20 mm with conventional techniques or as ≥10 mm with spiral CT scan.

Exclusion Criteria:

* Patient has a platelet count of < 100,000/uL within 14 days before enrollment.
* Patient has an absolute neutrophil count of < 1500/uL within 14 days before enrollment.
* Patient has a calculated or measured creatinine clearance of <30 mL/minute within 14 days before enrollment.
* Patient has ³Grade 2 peripheral neuropathy within 14 days before enrollment.
* Myocardial infarction within 6 months prior to enrollment or has New York Hospital Association (NYHA) Class III or IV heart failure (see section 8.4), uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at Screening has to be documented by the investigator as not medically relevant.
* Patient has hypersensitivity to bortezomib, boron or mannitol.
* Female subject is pregnant or breast-feeding. Confirmation that the subject is not pregnant must be established by a negative serum b-human chorionic gonadotropin (b-hCG) pregnancy test result obtained during screening. Pregnancy testing is not required for post-menopausal or surgically sterilized women.
* Patient has received other investigational drugs with 14 days before enrollment
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Patient has a cardiac ejection fraction < 50% by echocardiogram or MUGA scan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2006-07; Primary Completion 2007-11 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
To evaluate the rate of complete response to therapy defined as resolution of PET avidity in all previously documented sites at the completion of chemotherapy. | 1 year

SECONDARY OUTCOMES:
Assess toxicity | 1 year
evaluate event-free survival at 2 years | 2 years
evaluate overall survival at 2 years | 2 years
assess early PET restaging after 3 cycles of chemotherapy. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ann LaCasce, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States